CLINICAL TRIAL: NCT01261962
Title: Modulation of Immune Response by Oral Zinc Supplementation in Adjuvant Chemotherapy for Colon Cancer: a Study of Global Gene Expression and Function of Humoral Immunity and Neutrophils
Brief Title: Modulation of Immune Response by Oral Zinc Supplementation in Chemotherapy for Colon Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Selma Freire de Carvalho da Cunha, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FAPESP:2010/08787-1
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Adjuvant Chemotherapy; Colon Cancer; Immunity
Keywords: Humoral immunity; Neutrophil function; Gene expression
MeSH Terms: conditions — Colonic Neoplasms | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Chemotherapy and zinc (Experimental): Patients in adjuvant chemotherapy supplemented with zinc
  Interventions: Dietary Supplement: zinc
- Chemotherapy placebo (Placebo Comparator): Patients in adjuvant chemotherapy with placebo
  Interventions: Other: Placebo
- Control and zinc (Other): Healthy patients supplemented with zinc
  Interventions: Dietary Supplement: zinc
- Control Placebo (Other): Healthy volunteers received placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: zinc — zinc sulfate, 35 mg twice daily for 4 months
  Arms: Chemotherapy and zinc; Control and zinc
Other: Placebo — Placebo, One capsule, twice daily for 4 months
  Arms: Chemotherapy placebo; Control Placebo

SUMMARY:
In leukocytes of patients undergoing adjuvant chemotherapy for colon cancer treatment: a)identify genes modulated by oral supplementation of zinc; b) evaluate the effects of oral zinc supplementation on humoral immunity and neutrophil function. The study will be conducted on 30 adult patients aged grater than 18 years, of both genders who have undergone surgical resection of colonic neoplastic lesions without metastatic lesion. Patients will be randomized into two groups, with the first (Group QT Zn, n = 15) receive 70 mg/d of zinc for 16 weeks and the second will receive placebo (QT Placebo Group, n = 15). The study will also include 30 healthy volunteers who receive supplementation of 70 mg/d of Zn (C Zn group, n = 15) or placebo (Group C Placebo, n = 15). Zinc supplementation or placebo for all study groups will start two days before the volunteers received the pneumococcal vaccine, polyvalent 23. Fifteen days after vaccination, patients begin chemotherapy as pre-established criteria by the Oncology Service. Will be monitored the parameters of nutritional status (anthropometry, bioelectrical impedance, food intake, and laboratory tests) adverse effects, according to rules of the CTCAE. In the evaluation of humoral immunity, antibodies opsonization and in the pneumococcal polysaccharide will be measured. Will be evaluated the function of neutrophils by measuring DNA NETs and quantified calprotectin and elastase released in the culture supernatants of activated neutrophils. RT-qPCR will be done of genes differentially expressed(DEGS) on activated leukocytes. In six volunteers from each group will be analyzed global gene expression from RNA extracted from leukocytes by microarray; will be detected and correlated the molecular pathways modulated by zinc by MetaCore software (GeneGo). The DEGS will be validated by RT-qPCR.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Diagnostic histopathology of colon cancer stage III (Dukes' stage C)
* Performance Scale Karnofsky greater or equal to 70%
* Have been subjected to resection of the primary neoplastic lesion in more than 8 weeks before start of chemotherapy
* Patient in the first cycle of chemotherapy in adjuvant XELOX regimen.

Exclusion Criteria:

* Patients with a history of autoimmune or inflammatory disease, active infectious disease, liver disease, renal failure or diabetes mellitus
* Patients with metastatic disease
* Have previously received radiotherapy or chemotherapy
* Use of GCSF-Granulokine ® (growth-stimulating factor granulocyte)
* Use of immunosuppressive drugs, diuretics and supplements of zinc or copper.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-12 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Gene expression | 18 months
  Modulation of genes related to immune response

SECONDARY OUTCOMES:
Humoral immunity and neutrophil function | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Selma Freire C. Cunha, PhD, Study Director — Sao Paulo University; Camila Bitu M. Braga, Msc, Principal Investigator — Sao Paulo University
Locations (1):
- Departament of Clinical Oncology, Sao Paulo University, Ribeirão Preto, São Paulo, Brazil